CLINICAL TRIAL: NCT03269474
Title: Computational Drug Repurposing for All Epidermolysis Bullosa Simplex (EBS) Cases
Brief Title: Computational Drug Repurposing for All EBS Cases
Status: Recruiting | Type: Observational
Sponsor: Joyce Teng (Other)
Responsible Party: Sponsor-Investigator, Joyce Teng, Director of Pediatric Dermatology, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 41142
Record Dates: First submitted 2017-08-21; First posted 2017-08-31 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Epidermolysis Bullosa; Healthy; Genetic Skin Disease; Epidermolysis Bullosa Simplex; Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica
Keywords: epidermolysis bullosa; genetic expression; drug repurposing; computational approaches; drug discovery
MeSH Terms: conditions — Epidermolysis Bullosa; Skin Diseases, Genetic; Epidermolysis Bullosa Simplex; Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Punch biopsies of non-blistering and blistering skin, and peripheral blood mononuclear cells (PBMCs): CD8+ cytotoxic T cells and CD4+ helper T cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Blood and tissue specimen will be collected from subjects with an EB diagnosis. Tissue specimen will be collected from blistered and nonblistered skin.
  Interventions: Procedure: Experimental Group
- Control Group: Blood and tissue specimen will be collected from healthy subjects with non-EB. Tissue specimen will be collected from an inconspicuous skin area.
  Interventions: Procedure: Experimental Group

INTERVENTIONS:
Procedure: Experimental Group — Subjects with EB diagnosis

SUMMARY:
The study will compare gene expression differences between blistered and non-blistered skin from individuals with all subtypes of EB, as well as normal skin from non-EB subjects. State of the art computational analysis will be performed to help identify new drugs that might help all EB wound healing and reduce pain. Researchers will focus on drugs that have already been approved for treatment of other dermatologic or non-dermatologic diseases, and therefore be repurposed for treatment of EB. Drug development is a very expensive process taking decades for execution. Drug repurposing on the other hand, significantly reduces the cost and shortens the amount of time that is needed to bring effective treatments to clinical use. To date, there is no specific treatment targeting the physiology and immunologic response in EB patients during wound healing. Market availability of repurposed medications will provide all EB patients rapid access to treatments, thus improving their quality of life.

DETAILED DESCRIPTION:
Although gene, cell, and protein-based therapies are in development for patients suffering from all subtypes of epidermolysis bullosa (EB), new pharmacological treatments are in dire need. Characterizing molecular changes in EB, including gene expression, can identify new therapeutic targets and drugs that modulate those targets. However, sifting through gene expression information to identify the most promising drug targets is a complex data challenge. The goal of the study will identify a computational approach to evaluate and identify existing drugs approved for other diseases that can be repurposed for EB patients. The study will perform an unprecedented characterization of gene expression changes in EB patients compared to healthy, non-EB individuals across multiple tissues. Using a validated computational drug discovery platform, researchers will analyze gene expression and drug data using unique algorithms. In the first year, a list of ten, safety drugs more probable to treat the EB disease state will be identified. The most promising drugs discovered will then be tested in the clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of all ages
* Diagnosis of all subtypes of EB subjects
* Healthy, non-EB subjects
* Ability to complete study visit to collect tissue and blood specimen

Exclusion Criteria:

* Pregnancy, breast feeding
* Prior history of liver disease
* Serious known concurrent medical illness or infection, which could potentially present a safety risk and/or prevent tissue collection from subjects

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subject of all ages with either 1) a diagnosis of EB subjects or 2) healthy, non-EB subjects
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize gene expression changes in EB using RNA sequencing (RNA-seq) and Computational Profiling Potential Drug Targets | Through the completion of study in 1 year.
  Using bioinformatic algorithms to identify changes in gene expression and review of over 2000 FDA-approved drugs based on predicted modulation of gene expression changes using a computational evolutionary algorithm system.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce M Teng, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Pediatric Dermatology Clinic at Stanford Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
As of now, there are no plans to share the data with other researchers. Once the outcome measures have been accomplished, the research team will publish results for the entire clinicaltrials.gov community and researchers for this vulnerable population study.

REFERENCES:
- [Background] McLaren PJ, Mayne M, Rosser S, Moffatt T, Becker KG, Plummer FA, Fowke KR. Antigen-specific gene expression profiles of peripheral blood mononuclear cells do not reflect those of T-lymphocyte subsets. Clin Diagn Lab Immunol. 2004 Sep;11(5):977-82. doi: 10.1128/CDLI.11.5.977-982.2004. PMID 15358662
- [Background] Sleasman JW, Leon BH, Aleixo LF, Rojas M, Goodenow MM. Immunomagnetic selection of purified monocyte and lymphocyte populations from peripheral blood mononuclear cells following cryopreservation. Clin Diagn Lab Immunol. 1997 Nov;4(6):653-8. doi: 10.1128/cdli.4.6.653-658.1997. PMID 9384284
- [Background] Bray NL, Pimentel H, Melsted P, Pachter L. Near-optimal probabilistic RNA-seq quantification. Nat Biotechnol. 2016 May;34(5):525-7. doi: 10.1038/nbt.3519. Epub 2016 Apr 4. PMID 27043002
- [Background] Robinson MD, McCarthy DJ, Smyth GK. edgeR: a Bioconductor package for differential expression analysis of digital gene expression data. Bioinformatics. 2010 Jan 1;26(1):139-40. doi: 10.1093/bioinformatics/btp616. Epub 2009 Nov 11. PMID 19910308
- [Background] Law V, Knox C, Djoumbou Y, Jewison T, Guo AC, Liu Y, Maciejewski A, Arndt D, Wilson M, Neveu V, Tang A, Gabriel G, Ly C, Adamjee S, Dame ZT, Han B, Zhou Y, Wishart DS. DrugBank 4.0: shedding new light on drug metabolism. Nucleic Acids Res. 2014 Jan;42(Database issue):D1091-7. doi: 10.1093/nar/gkt1068. Epub 2013 Nov 6. PMID 24203711
- [Background] Sugaya N, Kanai S, Furuya T. Dr. PIAS 2.0: an update of a database of predicted druggable protein-protein interactions. Database (Oxford). 2012 Oct 10;2012:bas034. doi: 10.1093/database/bas034. Print 2012. PMID 23060433
- [Background] Subramanian A, Kuehn H, Gould J, Tamayo P, Mesirov JP. GSEA-P: a desktop application for Gene Set Enrichment Analysis. Bioinformatics. 2007 Dec 1;23(23):3251-3. doi: 10.1093/bioinformatics/btm369. Epub 2007 Jul 20. PMID 17644558
- [Result] Cohn HI, Teng JM. Advancement in management of epidermolysis bullosa. Curr Opin Pediatr. 2016 Aug;28(4):507-16. doi: 10.1097/MOP.0000000000000380. PMID 27386970
- [Result] Uitto J, Bruckner-Tuderman L, Christiano AM, McGrath JA, Has C, South AP, Kopelan B, Robinson EC. Progress toward Treatment and Cure of Epidermolysis Bullosa: Summary of the DEBRA International Research Symposium EB2015. J Invest Dermatol. 2016 Feb;136(2):352-358. doi: 10.1016/j.jid.2015.10.050. PMID 26802230
- [Result] Nystrom A, Thriene K, Mittapalli V, Kern JS, Kiritsi D, Dengjel J, Bruckner-Tuderman L. Losartan ameliorates dystrophic epidermolysis bullosa and uncovers new disease mechanisms. EMBO Mol Med. 2015 Sep;7(9):1211-28. doi: 10.15252/emmm.201505061. PMID 26194911
- [Result] Wally V, Kitzmueller S, Lagler F, Moder A, Hitzl W, Wolkersdorfer M, Hofbauer P, Felder TK, Dornauer M, Diem A, Eiler N, Bauer JW. Topical diacerein for epidermolysis bullosa: a randomized controlled pilot study. Orphanet J Rare Dis. 2013 May 7;8:69. doi: 10.1186/1750-1172-8-69. PMID 23651789
- [Result] Li J, Zheng S, Chen B, Butte AJ, Swamidass SJ, Lu Z. A survey of current trends in computational drug repositioning. Brief Bioinform. 2016 Jan;17(1):2-12. doi: 10.1093/bib/bbv020. Epub 2015 Mar 31. PMID 25832646
- [Result] Low YS, Daugherty AC, Schroeder EA, Chen W, Seto T, Weber S, Lim M, Hastie T, Mathur M, Desai M, Farrington C, Radin AA, Sirota M, Kenkare P, Thompson CA, Yu PP, Gomez SL, Sledge GW Jr, Kurian AW, Shah NH. Synergistic drug combinations from electronic health records and gene expression. J Am Med Inform Assoc. 2017 May 1;24(3):565-576. doi: 10.1093/jamia/ocw161. PMID 27940607
- [Result] Bchetnia M, Tremblay ML, Leclerc G, Duperee A, Powell J, McCuaig C, Morin C, Legendre-Guillemin V, Laprise C. Expression signature of epidermolysis bullosa simplex. Hum Genet. 2012 Mar;131(3):393-406. doi: 10.1007/s00439-011-1077-7. Epub 2011 Aug 30. PMID 21877134
- [Result] Roth W, Reuter U, Wohlenberg C, Bruckner-Tuderman L, Magin TM. Cytokines as genetic modifiers in K5-/- mice and in human epidermolysis bullosa simplex. Hum Mutat. 2009 May;30(5):832-41. doi: 10.1002/humu.20981. PMID 19267394
- [Result] Lee B, Geyfman M, Andersen B, Dai X. Analysis of gene expression in skin using laser capture microdissection. Methods Mol Biol. 2013;989:109-17. doi: 10.1007/978-1-62703-330-5_10. PMID 23483391
- [Result] Lovendorf MB, Mitsui H, Zibert JR, Ropke MA, Hafner M, Dyring-Andersen B, Bonefeld CM, Krueger JG, Skov L. Laser capture microdissection followed by next-generation sequencing identifies disease-related microRNAs in psoriatic skin that reflect systemic microRNA changes in psoriasis. Exp Dermatol. 2015 Mar;24(3):187-93. doi: 10.1111/exd.12604. PMID 25431026